CLINICAL TRIAL: NCT04894890
Title: A Prospective Multicenter Study for the Assessment of Treatment Patterns, Effectiveness and Safety of Secukinumab in Adult Patients With Moderate to Severe Plaque Psoriasis in a Real-world Setting in China
Acronym: UNMASK2
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457ACN06
Record Dates: First submitted 2021-05-18; First posted 2021-05-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis
Keywords: psoriasis; China; secukinumab; real world study
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- secukinumab: Patients administered secukinumab by prescription
  Interventions: Drug: secukinumab

INTERVENTIONS:
Drug: secukinumab — There is no treatment allocation. Patients administered secukinumab by prescription that have started before inclusion of the patient into the study will be enrolled.
  Other Names: Cosentyx

SUMMARY:
This non-interventional, prospective, multi-center study aims to provide short- and long- term treatment patterns, effectiveness, and safety of secukinumab in Chinese patients with moderate to severe plaque psoriasis (with and without PsA) initiating treatment of secukinumab.

DETAILED DESCRIPTION:
All patients will be followed up for 52 weeks no matter they adhere to secukinumab or they have shifted to other treatment plans. Data will be collected in conjunction with routine care visits, most likely happen at week 0, 4, 12, 16, 24, 36, 52. No extra study visits, examinations, laboratory tests or procedures will be mandated. If visits happen at other time points (not within the window period), then they will be counted as unscheduled visits.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years;
* Diagnosis of clinically moderate to severe plaque-psoriasis;
* Initiating treatment with secukinumab during the identification period or within 30 days prior to the index date;
* Patient agrees to sign the informed consent

Exclusion Criteria:

- Participation in any dermatology or rheumatology clinical trial, concurrent or within the last 30 days of the secukinumab initiating date

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed diagnosis of moderate to severe plaque psoriasis initiating secukinumab will be eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 1002 (Actual)
Dates: Start 2021-09-26 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving a 90% reduction in the Psoriasis Area and Severity Index (PASI) score | week 24
  The PASI is used for assessing and grading the severity of psoriatic lesions and their response to therapy. PASI scores can range from a lower value of 0, corresponding to no signs of psoriasis, up to a theoretic maximum of 72.0.

SECONDARY OUTCOMES:
Percentage of patients experiencing a 75% reduction of PASI (PASI75) | week 4, week12, week 16, week 24, week 36, week 52
  The PASI is used for assessing and grading the severity of psoriatic lesions and their response to therapy. PASI scores can range from a lower value of 0, corresponding to no signs of psoriasis, up to a theoretic maximum of 72.0.
Percentage of patients experiencing a 90% reduction of PASI (PASI90) | week 4, week12, week 16, week 36, week 52
  The PASI is used for assessing and grading the severity of psoriatic lesions and their response to therapy. PASI scores can range from a lower value of 0, corresponding to no signs of psoriasis, up to a theoretic maximum of 72.0.
Percentage of patients experiencing a 100% reduction of PASI (PASI100) | week 4, week12, week 16, week 24, week 36, week 52
  The PASI is used for assessing and grading the severity of psoriatic lesions and their response to therapy. PASI scores can range from a lower value of 0, corresponding to no signs of psoriasis, up to a theoretic maximum of 72.0.
Percentage of patients with absolute PASI change ≤1, ≤2, ≤3,and ≤5 | week 4, week12, week 16, week 24, week 36, week 52
  The PASI is used for assessing and grading the severity of psoriatic lesions and their response to therapy. PASI scores can range from a lower value of 0, corresponding to no signs of psoriasis, up to a theoretic maximum of 72.0
Percentage of patients with Investigator Global Assessment Mod 2011 (IGA mod 2011) 0 or 1 | week 4, week12, week 16, week 24, week 36, week 52
  The IGA mod 2011 rating scale for overall psoriatic disease can range from 0 to 4 (0: Clear, 1: almost clear, 2: mild, 3: moderate, 4: severe)
Mean change of Investigator Global Assessment Mod 2011(IGA mod 2011) | week 4, week12, week 16, week 24, week 36, week 52
  The IGA mod 2011 rating scale for overall psoriatic disease can range from 0 to 4 (0: Clear, 1: almost clear, 2: mild, 3: moderate, 4: severe)
Percentage of patients achieved (Body Surface Area) BSA≤1% | week 4, week12, week 16, week 24, week 36, week 52
  The total BSA affected by plaque-type psoriasis will be estimated from the percentages of areas affected, including head, trunk, upper limbs and lower limbs.
  The following calculations will be done: each reported percentage will be multiplied by its respective body region corresponding factor (head = 0.1, trunk = 0.3, upper limbs = 0.2, lower limbs = 0.4). The resulting four percentages will be added up to estimate the total BSA affected by psoriasis.
Mean change in Dermatology life quality index (DLQI) | Baseline,week 4, week12, week 16, week 24, week 36, week 52
  DLQI is a 10-item general dermatology disability index designed to assess HRQoL in adult patients with skin diseases such as eczema, psoriasis, acne and viral warts. The measure is self-administered and includes domains of daily activities, leisure, personal relationships, symptoms and feelings, treatment and work/school.
  Each item has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions.
  Scores range from 0 to 30 and higher scores indicate greater HRQoL impairment. Additionally, each subscale of the DLQI may be analyzed separately.
Percentage of patients achieving DLQI 0 or 1 response | week 4, week12, week 16, week 24, week 36, week 52
  DLQI is a 10-item general dermatology disability index designed to assess HRQoL in adult patients with skin diseases such as eczema, psoriasis, acne and viral warts. The measure is self-administered and includes domains of daily activities, leisure, personal relationships, symptoms and feelings, treatment and work/school.
  Each item has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions.
  Scores range from 0 to 30 and higher scores indicate greater HRQoL impairment. Additionally, each subscale of the DLQI may be analyzed separately.
Incidence of AEs/SAEs | 52 weeks
  An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
  Serious adverse event (SAE) is defined as an AE which results in death or is life-threatening, persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, requires inpatient hospitalization or prolongation of existing hospitalization or is medically significant
Incidence of treatment-related AEs on-treatment and post-discontinuation follow up | 52 weeks
  An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Incidence of unexpected treatment related AEs/SAEs on-treatment and post-discontinuation follow up | 52 weeks
  An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
  Serious adverse event (SAE) is defined as an AE which results in death or is life-threatening, persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, requires inpatient hospitalization or prolongation of existing hospitalization or is medically significant
Incidence of treatment-related SAEs on-treatment and post-discontinuation follow up | 52 weeks
  Serious adverse event (SAE) is defined as an AE which results in death or is life-threatening, persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, requires inpatient hospitalization or prolongation of existing hospitalization or is medically significant
Incidence of AEs of special interest on-treatment and post discontinuation follow up | 52 weeks
  An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Proportion of patients experiencing at least one AE | 52 weeks
  An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Average number of AEs per patient | 52 weeks
  An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Percentage of secukinumab discontinuation caused by AE | 52 weeks
  An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Frequency distribution of patients by dosing pattern | 52 weeks
  Frequency distribution of patients by dosing pattern will be collected
Frequency distribution of patients by secukinumab retention | Week 4, week 12, week 16, week 24, week 36 and week 52
  Percentage of patients who are persistent secukinumab users or who discontinue secukinumab
Mean (SD) time to secukinumab discontinuation | Up to 52 weeks
  Mean (SD) time to secukinumab discontinuation will be collected
Median (interquartile range) time to secukinumab discontinuation | 52 weeks
  Median (IQR) time to secukinumab discontinuation will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (34):
- China (34):
  - Novartis Investigative Site, Xicheng Direct, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Lanzhou, Gansu
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Guangdong, Guangzhou
  - Novartis Investigative Site, Haikou, Hainan
  - Novartis Investigative Site, Handan, Hebei
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Xuzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Yinchuan, Ningxia
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Qingdo, Shandong
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Nanjing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Shanyang
  - Novartis Investigative Site, Tianjin
  - Novartis Investigative Site, Wuhan
  - Novartis Investigative Site, Zhejiang

IPD SHARING:
Plan to Share IPD: No